CLINICAL TRIAL: NCT05307523
Title: Up and Down: Use of Dynamic Partial Body Weight Support Play Environment to Encourage Upright Mobility and Exploration in Infants With Down Syndrome (DS)
Brief Title: Use of Partial Body Weight Support Play Environment to Encourage Mobility and Exploration in Infants With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Heather Feldner, Assistant Professor, School of Medicine Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00014183
Record Dates: First submitted 2022-01-21; First posted 2022-04-01 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Down Syndrome; Trisomy 21
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: This pilot study uses a randomized, crossover design with children serving as their own controls. Study activities for each child will take place over 9 weeks. Children and their families will come to one of the research labs to participate, one family at a time. On the first visit, parents will be asked to review and sign an informed consent document to participate and baseline assessments will be completed. The intervention will take place during weeks 2-4 and weeks 6-8, with a washout and reassessment period during week 5 prior to crossover. A final reassessment session will take place during week 9.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Enriched Environment Play With Harness Support (Experimental): Enriched environment play, movement, and exploration for children with Down Syndrome while using a portable partial body weight support harness to facilitate movement and exploration.
  Interventions: Device: Enriched Play Environment with Partial Body Weight Support Harness
- Enriched Environment Play Without Harness Support (Active Comparator): Enriched environment play, movement, and exploration without additional partial body weight support provided.
  Interventions: Other: Enriched Play Environment without Partial Body Weight Support Harness

INTERVENTIONS:
Device: Enriched Play Environment with Partial Body Weight Support Harness — A low-tech portable canopy with a partial-body weight harness system that allows a child and their caregiver to play freely in an 81 square foot space, which provides partial body weight offset to support movement and exploration.
  Arms: Enriched Environment Play With Harness Support
Other: Enriched Play Environment without Partial Body Weight Support Harness — Child and caregiver will play freely in the 81 square foot play space without being connected to the partial body weight support harness.
  Arms: Enriched Environment Play Without Harness Support

SUMMARY:
To explore the effects of Partial Body Weight Support (PBWS) within an enriched play environment for infants with Down Syndrome (DS), who are not yet walking, to better understand how PWBS may impact their mobility; exploration; and overall activity level.

* Hypothesis1 A: Infants will demonstrate increased movement counts on an ActiGraph during intervention compared to a control phase. Hypothesis 1B: Infants will demonstrate a higher frequency of exploratory behaviors during the intervention as compared to a control phase.
* Hypothesis 2: Infants will demonstrate an increased rate of improvement in Gross Motor Function Measure scores after the intervention compared to a control phase.
* Hypothesis 3: Infants will demonstrate higher parent-reported mastery motivation on the Dimensions of Mastery Questionnaire after the intervention compared to a control phase.

DETAILED DESCRIPTION:
The procedures will take place within a portable play area, which includes toys and a partial body weight mobile harness system to assist the child in moving and exploring safely within the play area. Infants will always play and explore in this same area during the study but sometimes they will wear the PBWS harness and sometimes they will not wear the harness. During the intervention play sessions, the child will have the harness on. During the control play sessions, the child will play in the play area without the harness on. The child will participate in the intervention play sessions (using the harness) for 3 weeks, and in the control play sessions for 3 weeks. Before the first visit, this will be done randomly which group (intervention or control) the child will start with. Children will switch groups after week 5 of the study.

Week 1: assessment week, single session for 1 hour. At this first session, the investigators will do a developmental test for the child to see how they move around. This test will be videotaped. The investigators will also ask the caregiver to fill out a survey that asks caregivers questions about the motivation of their child and how they learn and play.

Week 2-4: play sessions, three times/week for one hour each. At each play session, the investigators will videotape the child playing and also place a small activity monitor on one wrist and one ankle. The session will end when the child has played in the play area for 30 minutes or the child has been present for 60 minutes, whichever comes first.

Week 5: assessment week, single session for 1 hour. The tests and surveys from the first week will be repeated. The child will then switch groups to or from the intervention group or the control group.

Weeks 6-8: play sessions, 3 times/week for one hour each. The child will participate in the same activities as described above but in the opposite group.

Week 9: assessment single session for 1 hour. The tests and surveys from week 1 and week 5 will be repeated a final time. The study will be over after this visit.

During all play and testing sessions, children will be given breaks as needed or if the caregiver request one. Caregivers will be able to play and interact with the child as they usually do throughout the play session and will be present in the play area with their children at all times.

ELIGIBILITY:
Inclusion Criteria:

* A medical diagnosis of DS (any form)
* Under 36 months old
* Able to sit independently
* One parent must be able to read proficiently enough in English to complete a written assessment.

Exclusion Criteria:

* The child is already taking independent steps
* The child has uncontrolled seizures
* The child has known medical precautions that would prohibit them from wearing a harness
* The child has other developmental disability diagnoses.

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-05-13 (Actual); Study Completion 2023-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Feldner, PT, PhD, PCS, Principal Investigator — University of Washingon
Locations (1):
- Center on Human Development and Disability (CHDD), Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data may be shared upon reasonable request to the research team.

REFERENCES:
- [Background] Campos JJ, Anderson DI, Barbu-Roth MA, Hubbard EM, Hertenstein MJ, Witherington D. Travel Broadens the Mind. Infancy. 2000 Apr;1(2):149-219. doi: 10.1207/S15327078IN0102_1. Epub 2000 Apr 1. PMID 32680291
- [Background] Lobo MA, Harbourne RT, Dusing SC, McCoy SW. Grounding early intervention: physical therapy cannot just be about motor skills anymore. Phys Ther. 2013 Jan;93(1):94-103. doi: 10.2522/ptj.20120158. Epub 2012 Sep 20. PMID 23001524
- [Background] Adolph KE, Hoch JE. Motor Development: Embodied, Embedded, Enculturated, and Enabling. Annu Rev Psychol. 2019 Jan 4;70:141-164. doi: 10.1146/annurev-psych-010418-102836. Epub 2018 Sep 26. PMID 30256718
- [Background] Waldman-Levi A, Erez AB. Will environmental interventions affect the level of mastery motivation among children with disabilities? A preliminary study. Occup Ther Int. 2015 Mar;22(1):19-27. doi: 10.1002/oti.1380. Epub 2014 Oct 13. PMID 25308165
- [Background] Kenyon LK, Farris JP, Aldrich NJ, Rhodes S. Does power mobility training impact a child's mastery motivation and spectrum of EEG activity? An exploratory project. Disabil Rehabil Assist Technol. 2018 Oct;13(7):665-673. doi: 10.1080/17483107.2017.1369587. Epub 2017 Aug 30. PMID 28853621
- [Background] Huang HH, Huang HW, Chen YM, Hsieh YH, Shih MK, Chen CL. Modified ride-on cars and mastery motivation in young children with disabilities: Effects of environmental modifications. Res Dev Disabil. 2018 Dec;83:37-46. doi: 10.1016/j.ridd.2018.08.001. Epub 2018 Aug 8. PMID 30098454
- [Background] Gilmore L, Cuskelly M. Associations of Child and Adolescent Mastery Motivation and Self-Regulation With Adult Outcomes: A Longitudinal Study of Individuals With Down Syndrome. Am J Intellect Dev Disabil. 2017 May;122(3):235-246. doi: 10.1352/1944-7558-122.3.235. PMID 28452583
- [Background] Glenn S, Dayus B, Cunningham C, Horgan M. Mastery motivation in children with Down syndrome. Downs Syndr Res Pract. 2001 Oct;7(2):52-9. doi: 10.3104/reports.114. PMID 11721530
- [Background] Almeida GL, Corcos DM, Latash ML. Practice and transfer effects during fast single-joint elbow movements in individuals with Down syndrome. Phys Ther. 1994 Nov;74(11):1000-12; discussion 1012-6. doi: 10.1093/ptj/74.11.1000. PMID 7972361
- [Background] Kokkoni E, Logan SW, Stoner T, Peffley T, Galloway JC. Use of an In-Home Body Weight Support System by a Child With Spina Bifida. Pediatr Phys Ther. 2018 Jul;30(3):E1-E6. doi: 10.1097/PEP.0000000000000516. PMID 29924078
- [Background] Kokkoni E, Mavroudi E, Zehfroosh A, Galloway JC, Vidal R, Heinz J, Tanner HG. GEARing smart environments for pediatric motor rehabilitation. J Neuroeng Rehabil. 2020 Feb 10;17(1):16. doi: 10.1186/s12984-020-0647-0. PMID 32041623
- [Derived] Abuatiq RA, Hoffman ME, LaForme Fiss A, Looper J, Feldner HA. Exploring the Efficacy of a Dynamic Harness System on Gross Motor Development and Motivation for Infants With Down Syndrome: A Pilot Study. Pediatr Phys Ther. 2024 Oct 1;36(4):468-476. doi: 10.1097/PEP.0000000000001130. Epub 2024 Oct 1. PMID 39073058

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on February 14, 2022, at a research office in the Center on Human Development and Disability (now called Institute on Human Development and Disability) and finished on May 13, 2023.
Pre-assignment Details: The initial assignment was random using the Excel randomization Function, then there was a washout period of one week after the first arm is completed
Groups:
- Group AB Enriched Environment Play (EEP) With Harness First: Enriched environment play, movement, and exploration for children with Down Syndrome while using a harness that provides portable partial body weight support to facilitate movement and exploration. This harness is a low-tech portable canopy with a partial-body weight harness system that allows a child and their caregiver to play freely in an 81-square-foot space and provides partial body weight offset to support movement and exploration.
  Then, Enriched Play Environment without the harness (Partial Body Weight Support).
  The child and caregiver will play freely in the 81-square-foot play space without being connected to the partial body weight support harness.
- Group BA Enriched Environment Play (EEP) Without Harness First: Enriched environment play, movement, and exploration for children with Down Syndrome while Not using the harness that provides a portable partial body weight support.
  Then, Enriched Play Environment with the use of the harness (Partial Body Weight Support). This harness is a low-tech portable canopy with a partial-body weight harness system that allows a child and their caregiver to play freely in an 81-square-foot space and provides partial body weight offset to support movement and exploration.
  The child and caregiver will play freely in the 81-square-foot play space without being connected to the partial body weight support harness.
Period: First Condition (3 Weeks)
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Started | 11 | 6
Completed | 9 | 6
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout (1 Week)
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Started (No interventions were administered during the washout. Re-assessment took place this week) | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0
Period: Second Condition (3 Weeks)
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Started | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group AB Enriched Environment Play (EEP) With Harness First: Enriched environment play, movement, and exploration for children with Down Syndrome while using a harness that provides portable partial body weight support to facilitate movement and exploration. This harness is a low-tech portable canopy with a partial-body weight harness system that allows a child and their caregiver to play freely in an 81-square-foot space and provides partial body weight offset to support movement and exploration.
  Then,Enriched Play Environment without the harness (Partial Body Weight Support).
  The child and caregiver will play freely in the 81-square-foot play space without being connected to the partial body weight support harness.
- Group BA Enriched Environment Play (EEP) Without Harness First: Enriched environment play, movement, and exploration for children with Down Syndrome while Not using the harness that provides a portable partial body weight support.
  Then, Enriched Play Environment with the use of the harness (Partial Body Weight Support). This harness is a low-tech portable canopy with a partial-body weight harness system that allows a child and their caregiver to play freely in an 81-square-foot space and provides partial body weight offset to support movement and exploration.
- Total: Total of all reporting groups
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: Months] | 19.10 (5.91) | 17.4 (6.56) | 18.39 (6.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 7 | 1 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 2 | 8
  White & Asian | 2 | 2 | 4
  American Indian or Alaska Native, White | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 6 | 17
Movement Counts Per 15 Seconds [Mean (Standard Deviation); unit: movement counts per 15 seconds] — Right Ankle mounted accelerometer (Actigraph GT3X+) data were collected at each assessment point. The sensors were placed on the child's right side ankle and covered with wristbands. The sensors were set to capture data in 1-second epochs during all play sessions. Mean activity counts were calculated by categorizing change in vector magnitude movement counts across a 15-second interval, with higher counts representing more lower extremity movement. Population: These measurements are excluding the 2 participants who dropped out of the AB group.
  movement counts per 15 seconds
    number analyzed (Participants) | 9 | 6 | 15
    (all) | 124.20 (99.99) | 227.21 (197.66) | 175.71 (148.83)
GMFM-88 [Mean (Standard Deviation); unit: Score on a scale] — The Gross Motor Function Measure-88 is a standardized, validated outcome measure in children with Down Syndrome used to assess progress in gross motor development domains of lying and rolling (score range 0-51), sitting (score range 0-60), crawling and kneeling (score range 0-42), standing (score range 0-39) and walking, running, and jumping (score range 0-72). Higher scores in each domain indicate better outcomes. Item scores are summed to calculate raw and percent scores for each of the five GMFM-88 dimensions. Dimension scores are averaged to obtain an overall total score. Population: These measurements exclude the 2 participants who dropped out of the AB group.
  Score on a scale
    number analyzed (Participants) | 9 | 6 | 15
    (all) | 45.7 (5.6) | 37.1 (11.5) | 41.4 (8.6)
DMQ-18 General Competency Scale [Mean (Standard Deviation); unit: score on a scale] — The Revised Dimensions of Mastery Questionnaire has one general competence scale and six mastery motivation scales of persistence: cognitive/object, gross motor, social-adults, social- children/peers, mastery pleasure, and negative reactions to challenge in mastery situations. It is completed by caregivers and has a score range of 41-205, with higher scores indicating greater mastery motivation observed for their child.
  The general competence score was calculated using the infant scoring formula [General Competence= Summing the scores of items 4+10+20+27+31, then the total is divided by 5. Population: These measurements are excluding the 2 participants who dropped out of the AB group.
  score on a scale
    number analyzed (Participants) | 9 | 6 | 15
    (all) | 1.8 (0.52) | 1.8 (0.61) | 1.8 (0.54)
Percentage of time spent upright [Mean (Standard Deviation); unit: percentage of time spent upright] — Percentage of time spent in upright positions (supported or unsupported standing, supported stepping, cruising), were assessed from R ankle-worn accelerometer data. Position was calculated using tri-axial orientation values of the accelerometer relative to the ground, and were verified using a behavioral video coding scheme that document child positioning every 6 seconds during a 30 minute play session. Percentage of time spent in each position was calculated at each assessment point, with higher percentages equating to more time spent upright and on feet. Population: These measurements do not include the 2 participants who dropped out of the AB group.
  percentage of time spent upright
    number analyzed (Participants) | 9 | 6 | 15
    (all) | 28.98 (19.63) | 23.44 (16.16) | 26.21 (17.90)

OUTCOME MEASURES:

1. Primary Outcome: Change in Movement Counts Per 15 Seconds From Baseline (Week 1) to Mid Study (Week 5)
Description: Right Ankle mounted accelerometer (Actigraph GT3X+) data were collected at each assessment point. The sensors were placed on the child's right side ankle and covered with wristbands. The sensors were set to capture data in 1-second epochs during all play sessions. Mean activity counts were calculated by categorizing change in vector magnitude movement counts across a 15-second interval, with higher counts representing more lower extremity movement.
Time Frame: Baseline (week 1) and mid study (week 5)
Population: 2 Dropped off
Measure: Mean (Standard Deviation); unit: movement counts per 15 seconds
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
movement counts per 15 seconds | -34.46 (66.93) | -88.62 (158.87)

2. Primary Outcome: Change in Movement Counts Per 15 Seconds From Mid Study (Week 5) to Final (Week 9)
Description: as for outcome 1
Time Frame: Mid study (week 5) and Final study (week 9)
Population: 2 dropped out
Measure: Mean (Standard Deviation); unit: movement counts per 15 seconds
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
movement counts per 15 seconds | 28.91 (61.49) | -9.75 (80.89)

3. Primary Outcome: Change in Movement Counts Per 15 Seconds From Baseline (Week 1) to Final (Week 9)
Description: as for outcome 1
Time Frame: Baseline (week 1) and Final Study (week 9)
Population: 2 dropped out
Measure: Mean (Standard Deviation); unit: movement counts per 15 seconds
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
movement counts per 15 seconds | 1.86 (68.99) | -98.75 (122.31)

4. Primary Outcome: Change in Gross Motor Performance Using the Gross Motor Function Measure-88 Scores From Baseline (Week 1) to Mid Study (Week 5)
Description: The Gross Motor Function Measure-88 is a standardized, validated outcome measure in children with Down Syndrome used to assess progress in gross motor development domains of lying and rolling (score range 0-51), sitting (score range 0-60), crawling and kneeling (score range 0-42), standing (score range 0-39) and walking, running, and jumping (score range 0-72). Higher scores in each domain indicate better outcomes. Item scores are summed to calculate raw and percent scores for each of the five GMFM-88 dimensions. Dimension scores are averaged to obtain an overall total score.
Time Frame: Baseline (week 1) and mid study (week 5)
Population: 2 dropped out
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
score on a scale | 7.01 (3.09) | 1.57 (2.89)
Statistical Analysis 1: Comparison: Group AB Enriched Environment Play (EEP) With Harness First vs Group BA Enriched Environment Play (EEP) Without Harness First; Test type: Other — Paired t-test for normally distributed data Wilcoxon Rank test for the not normally distributed data; p < 0.05, Both Paired T-test and Wilcoxon Rank — Paired T-test for the normally distributed data and a Wilcoxon Rank test for the non-parametric data were used; The data included both normally and not normally distributed data for the baseline, mid-study, and final study assessment points

5. Primary Outcome: Change in Gross Motor Performance Using the Gross Motor Function Measure-88 Scores From Mid Study (Week 5) to Final (Week 9)
Description: as for outcome 4
Time Frame: Mid study (Week 5) to Final (Week 9)
Population: 2 dropped out
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
score on a scale | 4.17 (2.85) | 6.28 (3.04)

6. Primary Outcome: Change in Gross Motor Performance Using the Gross Motor Function Measure-88 Scores From Baseline (Week 1) to Final (Weeks 9)
Description: as for outcome 4
Time Frame: Baseline (week 1) to Final study (week 9)
Population: 2 dropped out
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
score on a scale | 12.38 (3.84) | 8.81 (4.0)

7. Primary Outcome: Change in Caregiver Perception of Their Child's Mastery Motivation Using the Revised Dimensions of Mastery Questionnaire-18 Infant Version From Baseline (Week 1) to Mid Study (Week 5)
Description: The Revised Dimensions of Mastery Questionnaire has one general competence scale and six mastery motivation scales of persistence: cognitive/object, gross motor, social-adults, social- children/peers, mastery pleasure, and negative reactions to challenge in mastery situations. It is completed by caregivers and has a score range of 41-205, with higher scores indicating greater mastery motivation observed for their child.
  The general competence score was calculated using the infant scoring formula [General Competence= Summing the scores of items 4+10+20+27+31, then the total is divided by 5.
Time Frame: Baseline (week 1) and mid study (week 5)
Population: 2 dropped out
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
score on a scale | 0.47 (0.32) | 0.5 (0.52)

8. Primary Outcome: Change in Caregiver Perception of Their Child's Mastery Motivation Using the Revised Dimensions of Mastery Questionnaire-18 Infant Version From Mid Study (Week 5) to Final (Week 9)
Description: as for outcome 7
Time Frame: Mid study (week 5) to Final (week 9)
Population: 2 dropped out
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
score on a scale | 0.27 (0.35) | 0.43 (0.23)

9. Primary Outcome: Change in Caregiver Perception of Their Child's Mastery Motivation Using the Revised Dimensions of Mastery Questionnaire-18 Infant Version From Baseline (Week 1) to Final (Week 9)
Description: as for outcome 7
Time Frame: Baseline (week 1) to Final (week 9)
Population: 2 dropped out
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
score on a scale | 0.33 (0.32) | 0.67 (0.37)

10. Secondary Outcome: Change in Percentage of Time Spent in Upright (on Feet) Between Baseline (Week 1) and Mid Study (Week 5)
Description: Percentage of time spent in upright positions (supported or unsupported standing, supported stepping, cruising), were assessed from R ankle-worn accelerometer data. Position was calculated using tri-axial orientation values of the accelerometer relative to the ground, and were verified using a behavioral video coding scheme that document child positioning every 6 seconds during a 30 minute play session. Percentage of time spent in each position was calculated at each assessment point, with higher percentages equating to more time spent upright and on feet.
Time Frame: From baseline (week 1) to Mid study (week 5)
Population: 2 dropped out
Measure: Mean (Standard Deviation); unit: percentage of time spent in upright
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
percentage of time spent in upright | 9.61 (31.83) | -3.51 (15.1)

11. Secondary Outcome: Change in Percentage of Time Spent in Upright (on Feet) Between Mid Study (Week 5) and Final (Week 9)
Description: as for outcome 10
Time Frame: Mid Study (week 5) to Final (week 9)
Population: 2 dropped out
Measure: Mean (Standard Deviation); unit: percentage of time spent in upright
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
percentage of time spent in upright | 1.7 (15.7) | 5.8 (28.6)

12. Secondary Outcome: Change in Percentage of Time Spent in Upright (on Feet) Between Baseline (Week 1) and Final Study (Week 9)
Description: as for outcome 10
Time Frame: Baseline (week 1) and Final Study (week 9)
Population: 2 dropped out
Measure: Mean (Standard Deviation); unit: percentage of time spent in upright
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness First | Group BA Enriched Environment Play (EEP) Without Harness First
Number analyzed (Participants) | 9 | 6
percentage of time spent in upright | 14.9 (20.8) | 3.56 (23.3)

ADVERSE EVENTS:
Time Frame: 9 weeks for each participant
Description: All the participants were clinically stable
Groups:
- Group AB Enriched Environment Play (EEP) With Harness: Enriched environment play, movement, and exploration for children with Down Syndrome while using a harness that provides portable partial body weight support to facilitate movement and exploration. This harness is a low-tech portable canopy with a partial-body weight harness system that allows a child and their caregiver to play freely in an 81-square-foot space and provides partial body weight offset to support movement and exploration.
- Group BA Enriched Environment Play (EEP) Without Harness: Enriched environment play, movement, and exploration for children with Down Syndrome while Not using the harness that provides a portable partial body weight support.
  The child and caregiver will play freely in the 81-square-foot play space without being connected to the partial body weight support harness.
Arm/Group | Group AB Enriched Environment Play (EEP) With Harness | Group BA Enriched Environment Play (EEP) Without Harness
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT05307523/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT05307523/SAP_001.pdf
  • Informed Consent Form (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT05307523/ICF_002.pdf